CLINICAL TRIAL: NCT03080792
Title: Pre-Exercise for Allogeneic Stem Cell Transplant Patients: a Pilot Study
Brief Title: Pre-Exercise for Allogeneic Stem Cell Transplant Patients
Acronym: PRESENT-P
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficult
Sponsor: University Hospital Heidelberg (Other)
Collaborators: University Hospital Freiburg (Other); University of Cologne (Other); University Hospital Dresden (Other)
Responsible Party: Principal Investigator, Joachim Wiskemann, PI, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PRESENT-P/ S-030/2016
Record Dates: First submitted 2016-12-16; First posted 2017-03-15 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Cancer, Hematological
Keywords: stem cell transplantation; exercise; high intensity interval training; resistance training; physical fitness; cancer
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Experimental): Exercise Intervention, moderate to high-intensity endurance and resistance exercise
  Interventions: Behavioral: Experimental: moderate to high-intensity exercise

INTERVENTIONS:
Behavioral: Experimental: moderate to high-intensity exercise — 2x per week endurance exercise (continuous moderate and high intensity intervall training on a cycle ergometer) and progressive resistance training (machine based hypertrophy training)

SUMMARY:
The PRESENT-P study is a one-arm exercise intervention study for hematological cancer patients prior allogeneic stem cell transplantation (allo-HCT). This pilot study will investigate in a prehabilitation approach the safety and feasibility of high-intensity exercise program directly prior transplantation.

DETAILED DESCRIPTION:
The major objective of PRESENT-P is to investigate the feasibility and safety of a high intensity endurance exercise training (HIIT) and progressive resistance exercise prior allo-HCT. This multicenter pilot study will include n=30 patients. Patients perform two supervised exercise sessions per week. Recruitment take place 6-12 weeks prior allogeneic stem cell transplantation. Further aims of this pilot study are: to estimate the number of eligible patients, evaluate the recruitment procedure, and to explore the effect of HIIT prior allo-HCT on maximal oxygen uptake (VO2peak),submaximal endurance capacity, muscle strength, patient-reported-outcomes including QoL and physical functioning.

ELIGIBILITY:
Inclusion Criteria:

* Hematological cancer, e.g. AML, CLL, MM
* Scheduled for allo-HCT at the University Clinic Heidelberg or other cooperation sites within the next 4-12 weeks
* Patients ≥ 18 years of age
* Sufficient German language skills
* Willing/ able to train at the provided exercise facilities twice per week and to take part in the scheduled testing
* Signed informed consent

Exclusion Criteria:

* Heart insufficiency > NYHA III or uncertain arrhythmia
* Uncontrolled hypertension
* Severe renal dysfunction (GFR < 30%, Creatinine> 3mg/dl)
* Reduced standing or walking ability
* Insufficient hematological capacity (either hemoglobin value below 8 g/dl or thrombocytes below 30.000/µL)
* Any other comorbidities that preclude participation in the exercise programs
* Engaging in systematic intense exercise training (at least 1h twice per week)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of supervised high-intensity aerobic exercise training and high-intensity resistance training prior allo-HCT in hematological cancer patients. Measured as adherence to the training protocol | 4-12 weeks
  Adherence is defined as >50% of prescribed exercise sessions completed.
Safety of supervised high-intensity exercise aerobic exercise training and high-intensity resistance training prior allo-HCT in hematological cancer | 4-12 weeks
  Minor and Major adverse events that are related to the exercise intervention

SECONDARY OUTCOMES:
Change in maximal oxygen uptake (VO2peak), assessed in a maximal incremental exercise test (CPET) on a cycle ergometer | 4-12 weeks
Change in submaximal endurance performance, assessed in a 6-minute walk test (6MWT) | 4-12 weeks
Change in maximal voluntary isometric contraction (MVIC) in a stationary dynamometer test | 4-12 weeks
Change in maximal voluntary isometric hand-grip strength | 4-12 weeks
Change in Quality of Life (QoL) | 4-12 weeks
  European Research and Treatment in Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
Change in Fatigue | 4-12 weeks
  Multidimensional Fatigue Inventory, MFI 20
Change in depression | 4-12 weeks
  Center for Epidemiologic Studies Depression Scale, CES-D
Body Composition | 4-12 weeks
  Bioelectrical impendance analysis
Estimate the number of eligible patients | 12 month
Evaluation of recruitment procedures | 12 month
  Description of possible recruiting procedures in the ambulatory and stationary setting.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Wiskemann, Dr., Principal Investigator — Heidelberg University Hospital, National Center for Tumor Disease, Division of Medical Oncology, Working Group Exercise Oncology
Locations (5):
- Germany (5):
  - University of Colone, Cologne
  - University Hospital Carl Gustav Carus Dresden, Dresden
  - UCT Frankfurt / Hospital North-West, Frankfurt
  - Medical Center - University Freiburg, Freiburg im Breisgau
  - Heidelberg University Hospital, Heidelberg

IPD SHARING:
Plan to Share IPD: No